CLINICAL TRIAL: NCT02609230
Title: A Phase I Dose-Escalation Study of Onc201 Administered Every One or Three Weeks in Advanced Solid Tumors and Multiple Myeloma
Brief Title: A Dose-Escalation Study of Onc201 Administered Every One or Three Weeks in Advanced Solid Tumors and Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PH-077; 15-1009 (Other: Fox Chase Cancer Center)
Record Dates: First submitted 2015-11-10; First posted 2015-11-20 (Estimated); Last update posted 2021-06-04 (Actual); Status verified 2021-06

CONDITIONS: Advanced Solid Tumors; Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — TIC10 compound

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): For the first arm (A), dose escalation will use the following single patient dose-escalation cohorts based on 'Design 4' proposed by Simon and colleagues: 125, 250, and 500 mg. every 3 weeks.
  Interventions: Drug: ONC-201
- B (Experimental): Following completion of Arm A dose escalation, subsequent cohorts will be tested in a minimum of 3 patients, the Arm B dose cohort will consist of dose levels administered every week (planned dosing of 250, 375, 500 and 625 mg).
  Interventions: Drug: ONC-201

INTERVENTIONS:
Drug: ONC-201

SUMMARY:
This study will determine the maximum tolerated dose (MTD) and/or the recommended phase II dose (RP2D) of single agent ONC201 in patients with advanced solid tumors or multiple myeloma.

DETAILED DESCRIPTION:
This phase 1 study will determine the maximum tolerated dose (MTD) and/or recommended phase II dose (RP2D) of ONC201, when given as a single agent, to patients with advanced solid tumors or multiple myeloma, in two dose schedules including every 3 weeks and weekly. For the first arm (A), dose escalation will use the following single patient dose-escalation cohorts based on 'Design 4' proposed by Simon and colleagues: 125, 250, 500, and 625 mg. Following completion of Arm A dose escalation, subsequent cohorts will be tested in a minimum of 3 patients. The Arm B dose cohort will consist of dose levels administered once every one week (planned dosing of 250, 375, 500 and 625 mg). Dependent on PK and PD data, or emerging efficacy data, additional dose levels in Arm A or Arm B may be explored.

For Arm A, single patient cohorts will be used until the first instance of DLT or the second instance of grade 2 toxicity. Either occurrence will lead to immediate use of a modified 3+3 design and ~40% dose increments. Arm B will use a 3 + 3 design for all cohorts. It is anticipated that 16 - 48 evaluable patients in the dose escalation and an additional 17 patients in the expansion phase will be enrolled into this study over the course of 2 years. Patients will receive ONC201 in 3-week cycles until disease progression, unacceptable toxicity, or the patient discontinues for any other reason. The maximum duration of treatment will be 12 months unless it is determined that a patient would derive benefit from continued therapy beyond 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Solid tumor specific:

   * Patients must have a histologically/cytologically confirmed primary solid tumor
   * Radiographic or clinical evidence of advanced/metastatic malignant disease that is resistant to standard therapy or for which no standard therapy is available. Lesions may be measurable or non-measurable
2. Multiple myeloma specific:

   * Confirmed evidence of disease progression from immediately prior MM therapy or refractory to the immediately prior treatment
   * Measurable disease M protein component in serum (at least 0.5 g/dL) and/or urine (if present), (>=0.2 g excreted in a 24 hour collection sample).
   * Subjects with free light chain only disease are excluded
3. All previous therapies for cancer, including radiotherapy, major surgery and investigational therapies discontinued for ≥ 14 days (≥ 28 days for mitomycin C or nitrosoureas ) before Cycle 1 Day 1 (C1D1), and all acute effects of any prior therapy resolved to baseline severity or Grade ≤ 1 Common Terminology Criteria for Adverse Events (CTCAE v4.03), except alopecia or parameters defined in this eligibility list
4. Age ≥ 18 years
5. ECOG performance status ≤ 1
6. Adequate organ and marrow function as defined below:

   * Absolute neutrophil count ≥1,000/mm3 without growth factor use ≤ 7 days prior to C1D1
   * Platelets ≥75,000/mm3 without platelet transfusion ≤ 7 days prior to C1D1
   * Hemoglobin >8.0 mg/dL without red blood cell transfusion ≤ 7 days prior to C1D1
   * Total serum bilirubin <1.5 X upper limit of normal (ULN)
   * AST (SGOT)/ALT (SGPT) ≤2 X ULN; ≤ 5 X ULN if there is liver involvement secondary to tumor
   * Serum creatinine ≤ 1.5 X ULN (OR creatinine clearance ≥ 60 mL/min/1.73 m2)
   * Serum or urine pregnancy test (for females of childbearing potential) negative ≤7 days of starting treatment
7. Ability to understand and the willingness to sign a written informed consent document and comply with the study scheduled visits, treatment plans, laboratory tests and other procedures.
8. Female patients must be surgically sterile or be postmenopausal, or must agree to use effective contraception during the period of the trial and for at least 90 days after completion of treatment. Male patients must be surgically sterile or must agree to use effective contraception during the period of the trial and for at least 90 days after completion of treatment. The decision of effective contraception will be based on the judgment of the principal investigator or a designated associate.

Exclusion Criteria:

1. Patients with symptomatic brain metastases are excluded. Patients with asymptomatic and treated CNS metastases may participate in this trial. The patient must have completed any prior treatment for CNS metastases > 28 days prior to study entry including radiotherapy or surgery. Steroids for the treatment of brain metastasis are not permitted.
2. Active inflammatory gastrointestinal disease, chronic diarrhea (unless related to underlying malignancy or prior related treatment) or history of abdominal fistula, gastrointestinal perforation, peptic ulcer disease, or intra-abdominal abscess within 6 months prior to study enrollment. Gastroesophageal reflux disease under treatment with proton pump inhibitors is allowed.
3. Pregnancy or breast feeding
4. Current active treatment in another clinical study
5. Active bacterial, fungal or viral infection including hepatitis B (HBV), hepatitis C (HCV), requiring treatment with IV antibiotic, IV anti-fungal, or anti-viral.
6. Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness.
7. Multiple myeloma specific:

   * Active or prior plasma cell leukemia (defined as either 20% of peripheral WBC comprised of plasma/CD138+ cells or an absolute count of 2 x 10^9/L)
   * Solitary bone or solitary extramedullary plasmacytoma as the only evidence of plasma cell dyscrasia.
8. Subjects with serum calcium (corrected for albumin) ≥ 12 mg/dL
9. Any of the following in the previous 6 months: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident, transient ischemic attack or symptomatic pulmonary embolism.
10. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, or in the judgment of the investigator would make the patient inappropriate for entry into the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2015-11-05 (Actual); Primary Completion 2020-03 (Actual); Study Completion 2020-03-26 (Actual)

PRIMARY OUTCOMES:
Determine the maximum tolerated dose of ONC201 | At day 21 of Cycle 1 of therapy

SECONDARY OUTCOMES:
Peak Plasma Concentration of ONC201 | 0, 0.5, 2, 4, 6, 24, 48, 72, 168 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Olszanski, MD, Principal Investigator — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania, United States